CLINICAL TRIAL: NCT03986255
Title: Identifying Biomarkers and Changes in Cerebrospinal Fluid Collected Pre and Post Spinal Cord Stimulation: A Single Centre, Prospective, Exploratory Study in Subjects Suffering From Chronic Refractory Pain Conditions
Brief Title: Identifying Biomarkers and Changes in Cerebrospinal Fluid Collected Pre and Post Spinal Cord Stimulation in Subjects Suffering From Chronic Refractory Pain Conditions
Acronym: CSF-STIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early at the request of Sponsors.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSF-STIM v1.0 22/OCT/2018; CSF-STIM (Other: Guy's and St Thomas Hospital)
Record Dates: First submitted 2019-02-27; First posted 2019-06-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar Puncture (Experimental): Participants will undergo Lumbar puncture procedure
  Interventions: Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: Lumbar Puncture — The participant is placed lateral or sitting position. Fluoroscopy may be used to guide sampling. Full aseptic technique is used throughout.
  The skin is prepared with either 2% chlorhexidine/70% alcohol or iodine. 1% lidocaine is used for skin local anesthesia an entry point is identified, this may be done using fluoroscopy. This will be at the lowest intervertebral foramina interspace to minimize the risk of spinal cord injury. A small amount to head up tilt will be allowed to optimize CSF flow.
  Sampling is done using a "needle through needle" technique. An epidural needle is used to identify the epidural space using loss of resistance to saline technique. A spinal needle (26G) is then passed through the epidural needle into the subarachnoid space. Correct entry is noted once CSF is noted in the needle hub and 5 ml taken. This sample is then sent off for analysis.
  Once the CSF is sampled, the needle is removed and pressure applied to the skin entry point.

SUMMARY:
This is a single center exploratory study in subjects suffering from chronic refractory pain to identify cellular, molecular and protein biomarkers within cerebrospinal fluid (CSF).

The study aims to identify any form of correlation between biological content of CSF and pain/treatment success. The study population include individuals suffering from chronic pain which has not been effectively treated with pharmacological treatment, medical intervention or alternative non-invasive treatments who have been scheduled for spinal cord stimulation.

DETAILED DESCRIPTION:
This is a single centre exploratory study in individuals suffering from chronic refractory pain to identify cellular, molecular and protein biomarkers within cerebrospinal fluid (CSF).

The investigators aim to identify any form of correlation between biological content of CSF and pain/ spinal cord stimulator (SCS) therapy success. '

CSF will be sampled before and after SCS therapy, the samples will be analysed to explore and identify biomarkers that are potentially relevant to the chronic pain conditions

. All eligible participants who are enrolled in the study will undergo screening assessment. Specifically, assessments will include pain scores assessed by Visual Analogue Scale (VAS), quality of life as assessed by the EQ-5D, disability as assessed by the Oswestry Disability Index (ODI), quality of sleep as assessed by Pittsburgh Sleep Quality Index (PSQI), Pain sensation as assessed by Pain Map and neuropathic pain as assessed by Douleu Neuropathique 4 (DN4).

During trial implant participants will have CSF sample taken using lumbar puncture technique.

Following collection CSF sample will be analysed to Identify potential biomarkers.

All participants will return to the clinic 14 (± 7) days following the procedure to assess the outcome of their SCS trial and complete assessments which include Pain Map, Pain VAS, DN4 , PSQI , ODI , EQ-5D and Patients Global Impression of Change (PGIC).

Following this participants will be followed up for end of study visit. The second CSF sample will be taken at this visit using lumbar puncture technique. At this visit participants will further be asked to complete assessments including Pain Map, Pain VAS, DN4 , PSQI , ODI ,EQ-5D and PGIC.

ELIGIBILITY:
Inclusion Criteria:

1. Be capable of understanding and signing a written consent form
2. Subjects suffering from chronic neuropathic pain which has not been effectively managed with pharmacotherapy, medical interventions or alternative non-invasive treatments
3. Pain VAS score ≥ 5 on more than 3 days a week at least over three months.
4. Subjects deemed a suitable candidate receive spinal cord stimulator device as determined by a pain management specialist
5. No known contraindication to spinal cord stimulation
6. Does not have an active systemic or local infection

Exclusion Criteria:

1. Structural abnormalities of the spine at L2-L3 that may impact study procedure
2. Severe scoliosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Pain VAS | 6 Months
  Visual Analogue Scale (VAS) used to assess improvements in pain. It is a continuous scale comprised of a horizontal line which is 10 centimeters (100mm) in length, anchored by 2 verbal descriptors, one which is no pain and the other worst imaginable pain. Lower scores denote a better outcome.
  Participants will be asked to complete this questionnaires at baseline and follow up visits.
Pain Map | 6 Months
  A pain checklist with a list of anatomical locations from which the participants selects relevant sites to the site of his/her pain. It is used to assess location of pain.
  Participants will be asked to complete this questionnaires at baseline and follow up visits.
Oswestry Disability Index (ODI) | 6 Months
  A self completed questionnaire used to assess changes in disability and health. The participants checks the statements which most closely resembles their situation. The scores for all the questions are summed with lower scores denote no disability.
  Participants will be asked to complete this questionnaires at baseline and follow up visits.
Patient Global Impression of Change (PGIC) | 6 Months
  Questionnaire used to assess patient satisfaction
  Participants will be asked to complete this questionnaires at follow up visits.
  .
Douleur Neuropathique 4 (DN4) | 6 Months
  A clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient and 3 items based on the clinical examination. The questionnaire used to assess neuropathic pain
  Participants will be asked to complete this questionnaires at baseline and follow up visits.
EQ-5D-5L | 6 Months
  A self report questionnaire used to assess improvements in quality of life.
  Participants will be asked to complete this questionnaires at baseline and follow up visits.
Pittsburgh Sleep Quality Index (PSQI) | 6 Months
  A self report questionnaire that will used to assess improvements in sleep quality. The questionnaire consists of 19 items which measures several different aspects of sleep. Each item is weighted on a 0 - 3 interval scale, the overall score is calculated by totalling the seven component scores. Lower scores denote a healthier sleep quality
  Participants will be asked to complete this questionnaires at baseline and follow up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas Hospital, London, United Kingdom